CLINICAL TRIAL: NCT02859896
Title: An Open-Label, Randomized, Parallel Group Study to Assess the Safety and Efficacy of Hectorol® (Doxercalciferol Capsules) in Pediatric Patients With Chronic Kidney Disease Stages 3 and 4 With Secondary Hyperparathyroidism Not Yet on Dialysis
Brief Title: Safety and Efficacy of Hectorol in Pediatric Patients With Chronic Kidney Disease Stage 3 and 4 With Secondary Hyperparathyroidism Not Yet on Dialysis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was conducted to fulfill a post-marketing commitment (PMC).FDA acknowledged the fulfillment of this PMC.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14314; U1111-1178-4657 (Registry Identifier: ICTRP)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Secondary Hyperparathyroidism-Chronic Kidney Disease
MeSH Terms: interventions — 1 alpha-hydroxyergocalciferol; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hectorol (Experimental): Hectorol (Doxercalciferol) will be administered orally two to three times weekly dependent on patient age. A dose titration scheme is used to individualize the dose to the patient's iPTH management.
  Interventions: Drug: Doxercalciferol (GZ427397)
- Rocaltrol (Active Comparator): Rocaltrol (Calcitriol) will be administered orally seven days/week. A dose titration scheme is used to individualize the dose to the patient's iPTH management.
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Doxercalciferol (GZ427397) — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Hectorol
  Arms: Hectorol
Drug: Calcitriol — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Rocaltrol
  Arms: Rocaltrol

SUMMARY:
Primary Objective:

Evaluate the effect of Hectorol® capsules in reducing elevated levels of intact parathyroid hormone (iPTH).

Secondary Objectives:

* Evaluate the safety profile of Hectorol® capsules versus Rocaltrol® (calcitriol) capsules.
* Determine the pharmacokinetic profile of 1,25-dihydroxyvitamin D2 after administration of Hectorol®.

DETAILED DESCRIPTION:
The total study duration per patient will be approximately up to 28 weeks.

ELIGIBILITY:
Inclusion criteria :

* Male or female aged 5 to 18 years old.
* Weight ≥15 kg.
* Chronic kidney disease (CKD) Stage 3 or 4 not on dialysis, defined as glomerular filtration rate (GFR) between 15 and 59 mL/min/1.73m^2 (established by Schwartz equation) at Week -2 visit.
* Intact parathyroid hormone (iPTH) value >100 pg/mL for CKD Stage 3 or >160 pg/mL for CKD Stage 4, at Week -2 visit.
* Signed informed consent/assent form.

Exclusion criteria:

* The patient has a serum 25-hydroxyvitamin D level <30 ng/mL at screening.
* The patient has a corrected calcium ≥10 mg/dL at the Week -2 visit.
* The patient has a serum phosphorus >4.5 mg/dL for children 13 to 18 years of age; >5.8 mg/dL for children 5 to 12 years of age at the Week -2 visit.
* The patient is anticipated to require maintenance hemodialysis within 3 months.
* The patient used cinacalcet or vitamin D sterol therapies such as calcitriol, doxercalciferol, or paricalcitol within 14 days prior to the baseline visit.
* The patient has a history of, or active, symptomatic heart disease within 12 months prior to the baseline (Week 0) visit.
* The patient currently has a chronic gastrointestinal disease (ie, malabsorption, severe chronic diarrhea, chronic ulcerative colitis, or ileostomy).
* The patient currently has primary hyperparathyroidism or has had a total parathyroidectomy.
* The patient has an active malignancy.
* The patient is unable to swallow a capsule in size similar to the Hectorol® and Rocaltrol® capsules.
* The patient has a history of sensitivity or allergy to doxercalciferol, calcitriol or other vitamin D analogs.
* The patient currently uses aluminum or magnesium-based binders.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving two consecutive ≥30% reductions in iPTH | Baseline up to Week 12

SECONDARY OUTCOMES:
Percentage change from baseline in iPTH | Baseline, Week 12, Week 24
Number of hypercalcemia events (albumin corrected serum calcium >10.2 mg/dL) | Up to Weeks 12 and 24
Number of participants with adverse events | Baseline up to Week 24
Assessment of pharmacokinetic (PK) parameter: Serum 1,25-dihydroxyvitamin D2 concentration-time data | At Week -2, Baseline, and then within 24 hours of the most recent dose of Hectorol® at Weeks 2, 4, 6, 8 or 10 (whichever week is not used for serial PK assessment), and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (23):
- United States (21):
  - Children's Hospital Of Alabama Site Number : 8400022, Birmingham, Alabama
  - Cedars Sinai Medical Center Site Number : 8400033, Los Angeles, California
  - UC DAVIS Medical Center Site Number : 8400005, Sacramento, California
  - Yale University School of Medicine Site Number : 8400029, New Haven, Connecticut
  - University of Miami Site Number : 8400006, Miami, Florida
  - Nicklaus Children's Hospital Site Number : 8400008, Miami, Florida
  - Rush University Medical Center Site Number : 8400020, Chicago, Illinois
  - University of Minnesota Site Number : 8400014, Minneapolis, Minnesota
  - Hackensack University Site Number : 8400010, Hackensack, New Jersey
  - Goryeb Children's Hospital Site Number : 8400016, Morristown, New Jersey
  - Cohen Children's Medical Center of NY Site Number : 8400017, New Hyde Park, New York
  - Mount Sinai Medical Center Site Number : 8400007, New York, New York
  - Duke University Medical Center Site Number : 8400034, Durham, North Carolina
  - East Carolina University, Brody School of Medicine Site Number : 8400025, Greenville, North Carolina
  - Children's Hospital of Pittsburgh Site Number : 8400028, Pittsburgh, Pennsylvania
  - Greenville Hospital System Site Number : 8400027, Greenville, South Carolina
  - Vanderbilt University Medical Center Site Number : 8400024, Nashville, Tennessee
  - Texas Children's Hospital Site Number : 8400013, Houston, Texas
  - University of Utah Site Number : 8400026, Salt Lake City, Utah
  - Virginia Commonwealth University Site Number : 8400009, Richmond, Virginia
  - Marshfield Clinic Site Number : 8400001, Marshfield, Wisconsin
- Chile (2):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Concepción, Región del Biobío

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org